CLINICAL TRIAL: NCT00684645
Title: Non-Interventional Study In Patients With Advanced And/Or Metastatic Renal Cell Carcinoma (mRCC) Treated With SUTENT®
Brief Title: Non-Interventional Study (NIS) In Patients With Advanced And/Or Metastatic Renal Cell Carcinoma (mRCC) Treated With SUTENT®
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A6181171
Record Dates: First submitted 2008-05-22; First posted 2008-05-26 (Estimated); Results first posted 2012-08-21 (Estimated); Last update posted 2012-08-21 (Estimated); Status verified 2012-07

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: Safety and tolerability of SUTENT® in patients with metastatic or advanced renal cell carcinoma after failure of cytokines in real-life setting.
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sunitinib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients treated with SUTENT®: Patients with metastatic or advanced renal cell carcinoma after failure of cytokines therapy.
  Interventions: Drug: SUTENT

INTERVENTIONS:
Drug: SUTENT — SUTENT® hard gelatin capsules containing 12.5 mg, 25 mg or 50 mg equivalent of sunitinib malate; daily dosage of 50 mg for 4 consecutive weeks followed by a 2-week rest period. Sutent is administered until disease progression or occurrence of unacceptable toxicity.

SUMMARY:
Primary objective: to increase knowledge about safety, tolerability, quality of life and efficacy under conditions of routine use of SUTENT®. Secondary objectives: treatment response, hypothyroidism prevalence.The efficacy will be assessed using the Objective Response Rate, Time to Progression based on the RECIST criteria and the ECOG performance data.

DETAILED DESCRIPTION:
180 patients will be enrolled at 20 key oncological centres, the sample size is sufficient for exploratory analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced or metastatic renal cell carcinoma.

Exclusion Criteria:

* No previous cytokines therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic and/or advanced renal cell carcinoma after failure of cytokines therapy.
Sampling Method: Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2008-06; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (14):
- Czechia (14):
  - Pfizer Investigational Site, Brno
  - Pfizer Investigational Site, Chomutov
  - Pfizer Investigational Site, České Budějovice
  - Pfizer Investigational Site, Fryštát
  - Pfizer Investigational Site, Hradec Králové
  - Pfizer Investigational Site, Jihlava
  - Pfizer Investigational Site, Liberec
  - Pfizer Investigational Site, Nová Ves pod Pleší
  - Pfizer Investigational Site, Nový Jičín
  - Pfizer Investigational Site, Ostrava
  - Pfizer Investigational Site, Pardubice
  - Pfizer Investigational Site, Pilsen
  - Pfizer Investigational Site, Prague
  - Pfizer Investigational Site, Zlín

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181171&StudyName=Non-Interventional%20Study%20%28NIS%29%20In%20Patients%20With%20Advanced%20And/Or%20Metastatic%20Renal%20Cell%20Carcinoma%20%28mRCC%29%20Treated%20With%20SUTENT%AE

RESULTS

PARTICIPANT FLOW:
Groups:
- Sunitinib: The use and dosage recommendations for Sunitinib (Sutent) were in accordance with the local Summary of Product Characteristics.
Period: Overall Study
Arm/Group | Sunitinib
Started | 186
Completed | 72
Not Completed | 114
Not completed — Death | 2
Not completed — Progressive disease | 67
Not completed — Adverse Event | 27
Not completed — Lost to Follow-up | 3
Not completed — Other | 15

BASELINE CHARACTERISTICS:
Arm/Group | Sunitinib
Number analyzed (Participants) | 186
Age, Customized [Number; unit: participants]
  18 to 44 years | 10
  45 to 64 years | 99
  65 years or more | 77
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58
  Male | 128
Involvement of Regional Lymph Nodes [Number; unit: participants] — The sum of participants may not be equal to the number of participants beginning the study. A participant may be included in more than one category, or a participant may not be included in any category.
  participants
    Iliac | 31
    Paraaortal | 25
    Paracaval | 6
Previous Anti-Tumor Therapy [Number; unit: participants] — The sum of participants may not be equal to the number of participants beginning the study. A participant may be included in more than one category, or a participant may not be included in any category.
  participants
    Prior Radiotherapy | 152
    Prior Chemotherapy | 173
    Prior Hormonal Therapy | 180
    Prior Immunotherapy | 35
    Prior Cancer Surgeries | 8
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: percentage of participants] — ECOG criteria: 0: Fully active. 1: Ambulatory, carry out work of a light or sedentary nature. 2: Ambulatory, capable of all selfcare. 3: Capable of limited selfcare, confined to bed or chair more than 50% of waking hours. 4: Completely disabled, no selfcare, totally confined to bed or chair. 5: Dead.
  percentage of participants
    ECOG Performance Status 0 | 23
    ECOG Performance Status 1 | 72
    ECOG Performance Status 2 | 5
    ECOG Performance Status 3 | 0
    ECOG Performance Status 4 | 0
    ECOG Performance Status 5 | 0
Frequency of Involved Disease Sites [Number; unit: participants] — The sum of participants may not be equal to the number of participants beginning the study. A participant may be included in more than one category, or a participant may not be included in any category.
  participants
    Adrenal | 5
    Bone | 32
    Chest wall | 1
    Kidney | 26
    Liver | 20
    Lung | 88
    Lymph node | 7
    Lymph node - Mediastinum | 13
    Lymph node - Other | 4
    Lymph node - Retroperitoneal | 12
    Lymph node - Supraclavicular | 2
    Lymph node - Regional | 2
    Mediastinum | 3
    Other | 13
    Pancreas | 4
    Pelvis | 1
    Peritoneum | 7
    Pleura | 1
    Skin | 1
    Spleen | 1
Prevalence of hypothyroidism [Number; unit: participants] — At baseline, participants were considered hypothyroid if the investigator indicated they had hypothyroidism (yes/no) on the case report form (CRF). At subsequent visits, thyroid-stimulating hormone (TSH) and free thyroxine (FT4) levels were measured and hypothyroidism was defined as a TSH level greater than (>)5.0 milli-International Units per liter (mIU/L) at that visit.
  participants
    Hypothyroidism present | 15
    Hypothyroidism absent | 171
Prevalence of Hypertension [Number; unit: participants] — Hypertension was defined as blood pressure >140/90 millimeters of Mercury (mm Hg). At baseline, presence/absence of hypertension was recorded. If either the presence/absence of hypertension question or the blood pressure at Baseline indicated that the participant currently had hypertension, then the participant was considered to have hypertension at baseline. At subsequent visits, hypertension status was determined in terms of the blood pressure recorded at that visit.
  participants
    Hypertension present | 119
    Hypertension absent | 67

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Objective Response
Description: Percentage of participants with objective response based assessment of confirmed complete response (CR) or confirmed partial response (PR). CR is defined as the disappearance of all target lesions. PR is defined as at least 30% decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions.
Time Frame: 12 months
Population: Full analysis set (FAS): all participants who received at least one dose of the study medication.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 186
percentage of participants | 25.3 [19.2 to 32.1]

2. Primary Outcome: Progression-free Survival (PFS)
Description: The period from study entry until disease progression, death, or date of last contact.
Time Frame: Baseline to measured progressive disease (up to 12 months)
Population: FAS
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sunitinib
Number analyzed (Participants) | 186
months | 9.8 [9.1 to 12.5]

3. Primary Outcome: Overall Survival (OS)
Description: OS is the duration from enrollment to death.
Time Frame: Baseline to date of death (up to 12 months)
Population: FAS
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Sunitinib
Number analyzed (Participants) | 186
months | NA [NA to NA] — NA=not available. No median available, very few deaths observed.

4. Primary Outcome: Percentage of Participants With Eastern Cooperative Oncology Group (ECOG) Performance Status at Week 6
Description: Following are ECOG grades. 0: Fully active, perform all pre-disease activities without restriction. 1: Restricted in physically strenuous activity but ambulatory, carry out work of a light or sedentary nature. 2: Ambulatory, capable of selfcare, unable to carry out any work activities, up and about more than (>) 50% of waking hours. 3: Capable of limited selfcare, confined to bed or chair >50% of waking hours. 4: Completely disabled, not capable of any selfcare, totally confined to bed or chair. 5: Dead. Participants in "Not reported" category were on study, had no data for this time point.
Time Frame: Week 6
Population: FAS. Percentages based on entire FAS population.
Measure: Number; unit: percentage of participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 186
percentage of participants
  ECOG Grade 0 | 18.8
  ECOG Grade 1 | 68.3
  ECOG Grade 2 | 8.6
  ECOG Grade 3 | 2.2
  ECOG Grade 4 | 0.0
  ECOG Grade 5 | 0.0
  Not Reported | 2.2

5. Primary Outcome: Percentage of Participants With Eastern Cooperative Oncology Group (ECOG) Performance Status at Month 3
Description: as for outcome 4
Time Frame: Month 3
Population: FAS. Percentages based on entire FAS population.
Measure: Number; unit: percentage of participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 186
percentage of participants
  ECOG Grade 0 | 16.7
  ECOG Grade 1 | 60.2
  ECOG Grade 2 | 10.2
  ECOG Grade 3 | 2.7
  ECOG Grade 4 | 0.0
  ECOG Grade 5 | 0.0
  Not Reported | 10.2

6. Primary Outcome: Percentage of Participants With Eastern Cooperative Oncology Group (ECOG) Performance Status at Month 6
Description: as for outcome 4
Time Frame: Month 6
Population: FAS. Percentages based on entire FAS population.
Measure: Number; unit: percentage of participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 186
percentage of participants
  ECOG Grade 0 | 14.5
  ECOG Grade 1 | 47.8
  ECOG Grade 2 | 4.3
  ECOG Grade 3 | 1.6
  ECOG Grade 4 | 1.1
  ECOG Grade 5 | 0.0
  Not Reported | 30.6

7. Primary Outcome: Percentage of Participants With Eastern Cooperative Oncology Group (ECOG) Performance Status at Month 9
Description: as for outcome 4
Time Frame: Month 9
Population: FAS. Percentages based on entire FAS population.
Measure: Number; unit: percentage of participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 186
percentage of participants
  ECOG Grade 0 | 11.8
  ECOG Grade 1 | 36.6
  ECOG Grade 2 | 4.8
  ECOG Grade 3 | 0.5
  ECOG Grade 4 | 0.0
  ECOG Grade 5 | 0.0
  Not Reported | 46.2

8. Primary Outcome: Percentage of Participants With Eastern Cooperative Oncology Group (ECOG) Performance Status at Month 12
Description: as for outcome 4
Time Frame: Month 12
Population: FAS. Percentages based on entire FAS population.
Measure: Number; unit: percentage of participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 186
percentage of participants
  ECOG Grade 0 | 15.1
  ECOG Grade 1 | 39.8
  ECOG Grade 2 | 8.1
  ECOG Grade 3 | 4.8
  ECOG Grade 4 | 0.5
  ECOG Grade 5 | 1.1
  Not Reported | 30.6

9. Primary Outcome: Correlation Between Sunitinib-induced Hypertension and Tumor Response to Treatment (PFS)
Description: Sunitinib-induced hypertension was determined using blood pressure recorded at each postbaseline visit. Once participants were identified as having sunitinib-induced hypertension, they retained that status at subsequent visits. PFS is the time from start of study treatment to first documentation of tumor response to treatment. Hazard ratio represents the relationship between sunitinib-induced hypertension and PFS (presence/absence of hypertension).
Time Frame: Baseline to date of first documentation of response to treatment (up to 12 months)
Population: FAS
Measure: Number; unit: participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 186
participants
  Sunitinib-induced hypertension starting at Week 6 | 39 [0.257 to 0.609]
  Sunitinib-induced hypertension starting at Month 3 | 16
  Sunitinib-induced hypertension starting at Month 6 | 11
  Sunitinib-induced hypertension starting at Month 9 | 12
  Sunitinib-induced hypertension starting Month 12 | 4
Statistical Analysis 1: Comparison: Sunitinib; Time to PFS was analyzed using survival analysis methodology. Model was fitted with sunitinib-induced hypertension included as a time-dependent covariate (presence versus absence of hypertension); Test type: Superiority or Other; p < 0.0001, Cox proportional hazard; Hazard Ratio (HR) = 0.395, 95% CI 2-sided [0.257 to 0.609]

10. Primary Outcome: Correlation Between Sunitinib-induced Hypertension and Tumor Response to Treatment (OS)
Description: Sunitinib-induced hypertension was determined using blood pressure recorded at each postbaseline visit. Once participants were identified as having sunitinib-induced hypertension, they retained that status at subsequent visits. OS is the time from start of study treatment to death. Hazard ratio represents the relationship between sunitinib-induced hypertension and OS.
Time Frame: Baseline to date of death (up to 12 months)
Population: FAS
Measure: Number; unit: participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 186
participants
  Sunitinib-induced hypertension starting at Week 6 | 39 [0.151 to 0.864]
  Sunitinib-induced hypertension starting at Month 3 | 16
  Sunitinib-induced hypertension starting at Month 6 | 11
  Sunitinib-induced hypertension starting at Month 9 | 12
  Sunitinib-induced hypertension starting Month 12 | 4
Statistical Analysis 1: Comparison: Sunitinib; Time to OS was analyzed using survival analysis methodology. Model was fitted with sunitinib-induced hypertension included as a time-dependent covariate (presence versus absence of hypertension); Test type: Superiority or Other; p = 0.0221, Cox proportional hazard; Hazard Ratio (HR) = 0.361, 95% CI 2-sided [0.151 to 0.864]

11. Primary Outcome: Percentage of Participants With Hypothyroidism
Description: TSH and FT4 levels were measured and hypothyroidism was defined as a TSH level >5.0 mIU/L at that time point.
Time Frame: Baseline, Months 3, 6, 9, 12
Population: FAS. n = number of participants with evaluable data at that time point.
Measure: Number; unit: percentage of participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 186
percentage of participants
  Baseline (n=186) | 8.1
  Month 3 (n=168) | 17.9
  Month 6 (n=131) | 18.3
  Month 9 (n=100) | 20.0
  Month 12 (n=134) | 20.9

12. Primary Outcome: Percentage of Participants With Hypertension
Description: Hypertension was defined as follows. Grade 1: Asymptomatic, transient (less than [<]24 hours) increase by >20mm Hg (diastolic) or to >150/100 mm Hg if previously within normal limits (WNL). Grade 2: Recurrent or persistent (24 hours or more) or symptomatic increase by >20 mm Hg (diastolic) or to >150/100 mm Hg if previously WNL. Grade 3: Requiring >1 drug or more intensive therapy than previously. Grade 4: Life-threatening. Grade 5: Death.
Time Frame: Baseline, Week 6, Months 3, 6, 9, 12
Population: FAS. n = number of participants with evaluable data at that time point.
Measure: Number; unit: percentage of participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 186
percentage of participants
  Baseline (n=186) | 64.0
  Week 6 (n=182) | 51.1
  Month 3 (n=168) | 48.8
  Month 6 (n=131) | 54.2
  Month 9 (n=100) | 54.0
  Month 12 (n=134) | 39.6

13. Other Pre Specified Outcome: Summary of Adverse Events for Participants Who Required Dose Modification
Description: Adverse events (AEs) or treatment-emergent adverse events (TEAEs) were defined as newly occurring or worsening after first dose. Study drug modifications included reduced dose or temporary discontinuation of treatment.
Time Frame: Baseline up to 12 months
Population: Number of participants analyzed = All participants who required dose modification because of an adverse event. The total number of participants may exceed the number of participants analyzed because one participant may have reported more than one adverse event.
Measure: Number; unit: participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 17
participants
  Anaemia | 2
  Leukopenia | 2
  Neutropenia | 1
  Thrombocytopenia | 6
  Hypothyroidism | 1
  Aphthous stomatitis | 1
  Stomatitis | 2
  Disease progression | 9
  Oedema peripheral | 1
  Pyrexia | 1
  Jaundice | 1
  Bronchopneumonia | 2
  Herpes dermatitis | 1
  Urinary tract infection | 2
  False positive investigation result | 1
  Decreased appetite | 2
  Osteonecrosis of jaw | 1
  Leukaemia | 1
  Renal cell carcinoma | 2
  Cerebellar syndrome | 1
  Cerebrovascular accident | 1
  Loss of consciousness | 1
  Haematuria | 1
  Renal disorder | 1
  Asthma | 1
  Haemoptysis | 1
  Pulmonary embolism | 1
  Dermatitis exfoliative | 1
  Palmar-plantar erythrodysaesthesia syndrome | 3
  Rash | 1
  Skin erosion | 1
  Swelling face | 1
  Deep vein thrombosis | 1
  Hypertension | 4
  Infarction | 1
  Venous thrombosis limb | 1

14. Other Pre Specified Outcome: Percentage of Participants With Treatment-emergent Hypertension, by Common Terminology Criteria for Adverse Events (CTCAE) Grade
Description: Sunitinib-induced hypertension: not present at baseline but developed through the study, or if present at baseline increased by more than (>) 20% during the study. Grade 1: Asymptomatic, transient (less than [<]24 hours) increase by >20 millimeters of Mercury (mm Hg) (diastolic) or to >150/100 mm Hg if previously within normal limits (WNL); Grade 2: Recurrent or persistent (>=24 hours) or symptomatic increase by >20 mm Hg (diastolic) or to >150/100 mm Hg if previously WNL; Grade 3: Requiring >1 drug or more intensive therapy than previously; Grade 4: Life-threatening; Grade 5: Death.
Time Frame: Baseline up to 12 months
Population: All participants
Measure: Number; unit: percentage of participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 186
percentage of participants
  Hypertension, Grade 1 | 3.2
  Hypertension, Grade 2 | 1.1
  Hypertension, Grade 3 | 0.5

15. Other Pre Specified Outcome: Percentage of Participants Responding to Treatment
Description: Response categories for target lesions: Complete response (CR): Disappearance of all target lesions; Partial response (PR): At least a 30% decrease in the sum of the longest dimensions, reference=baseline sum of longest dimensions; Progressive disease (PD): At least a 20% increase in the sum of the longest dimensions, or the appearance of 1 or more new lesions; Stable disease (SD): Not sufficient shrinkage to qualify for PR, not sufficient increase to qualify for PD; Reference for PD and SD: smallest sum of longest dimensions since treatment started.
Time Frame: 12 months
Population: All participants
Measure: Number; unit: percentage of participants
Arm/Group | Sunitinib
Number analyzed (Participants) | 186
percentage of participants
  Complete response | 2.2
  Partial response | 23.1
  Stable / No response | 46.2
  Progressive disease | 19.9

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Sunitinib
Serious Adverse Events (participants affected / at risk) | 31/186
Other Adverse Events (participants affected / at risk) | 52/186
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (N=186)
Anaemia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Cardiac failure (Cardiac disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Diverticulum intestinal (Gastrointestinal disorders) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 1
Disease progression (General disorders) | 15
Bronchopneumonia (Infections and infestations) | 1
Empyema (Infections and infestations) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Weight decreased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hypochloraemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Cerebellar syndrome (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Renal disorder (Renal and urinary disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Infarction (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib (N=186)
Anaemia (Blood and lymphatic system disorders) | 3
Leukopenia (Blood and lymphatic system disorders) | 3
Neutropenia (Blood and lymphatic system disorders) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 8
Hyperthyroidism (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 2
Aphthous stomatitis (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Duodenal ulcer (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Periodontitis (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 3
Adverse event (General disorders) | 1
Chest pain (General disorders) | 1
Disease progression (General disorders) | 1
Face oedema (General disorders) | 1
Fatigue (General disorders) | 4
Mucosal inflammation (General disorders) | 2
Oedema peripheral (General disorders) | 2
Pyrexia (General disorders) | 2
Jaundice (Hepatobiliary disorders) | 1
Bronchopneumonia (Infections and infestations) | 1
Herpes dermatitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Blood parathyroid hormone increased (Investigations) | 1
Blood thyroid stimulating hormone increased (Investigations) | 1
False positive investigation result (Investigations) | 1
Weight decreased (Investigations) | 2
Cachexia (Metabolism and nutrition disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Paraesthesia (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 4
Skin disorder (Skin and subcutaneous tissue disorders) | 1
Skin erosion (Skin and subcutaneous tissue disorders) | 1
Skin toxicity (Skin and subcutaneous tissue disorders) | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 8
Phlebitis (Vascular disorders) | 1
Varicose vein (Vascular disorders) | 1
Venous thrombosis limb (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.